CLINICAL TRIAL: NCT03063892
Title: Evaluating the Effect of Tranexamic Acid (TXA) on Reduction of Postoperative Blood Transfusion in Hip Fracture Patients
Brief Title: Effect of Tranexamic Acid (TXA) on Reduction of Postoperative Blood Transfusion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gregory M Georgiadis MD (Other)
Responsible Party: Sponsor-Investigator, Gregory M Georgiadis MD, Orthopedic Surgeon, ProMedica Health System
Organization: ProMedica Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GG082015
Record Dates: First submitted 2015-08-04; First posted 2017-02-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Placebo Comparator): Will receive intravenous Saline solution placebo bolus dose in the Emergency Center over 10 minutes. The subject will also receive intravenous Saline solution over 8 hours prior to surgery. Another dose will be administered at the time of incision and the final dose three hours later.
  Interventions: Drug: Saline solution
- Experimental Arm (Experimental): Will receive intravenous Tranexamic Acid (TXA) 15mg/kg (maximum 1 gram) bolus dose over 10 minutes in the Emergency Center. The subject will also receive an intravenous dose of Tranexamic Acid (TXA) 15mg/kg over 8 hours prior to surgery. Another 15mg/kg dose of Tranexamic Acid (TXA) will be administered over 10 minutes at the time of incision and the final dose (15mg/kg) of Tranexamic Acid (TXA) intravenously over 10 minutes three hours later.
  Interventions: Drug: Tranexamic Acid (TXA)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — Tranexamic acid is an antifibrinolytic used to control bleeding
  Other Names: Cyklokapron
  Arms: Experimental Arm
Drug: Saline solution — Saline solution is used as the placebo comparator
  Other Names: normal saline
  Arms: Control Arm

SUMMARY:
Tranexamic Acid (TXA) is an antifibrolytic medication used in total hip and knee arthroplasty to reduce the need for intraoperative and postoperative blood transfusions. Limited research is available on its use in hip fracture patients. We hypothesize that the use of TXA preoperatively, perioperatively, and postoperatively will decrease blood loss and need for blood transfusion postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 60 years
* Hip fracture requiring surgical intervention
* Signs consent and agrees to participate

Exclusion Criteria:

* Under the age of 60
* Does not sign consent or refuses participation
* Known hypersensitivity to tranexamic acid
* Multiple acute fractures
* Creatinine clearance <30
* History of seizures
* Active hormone therapy
* History of coagulation abnormality
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the last year or history or recurrent DVT/PE
* Myocardial infarction (MI) and/or stents within the past year
* History of intracranial hemorrhage
* Acquired defective color vision
* Patients admitted directly to nursing units or surgery without stay in the Emergency Center
* Patients who sustain fracture while hospitalized at ProMedica Toledo Hospital

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
proportion of patients requiring packed Red Blood Cell transfusion | 72 hours
  units, perioperative

SECONDARY OUTCOMES:
intraoperative blood loss | 24 hours
  mL
postoperative anemia | 72 hours
  Hgb <7g/dL

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Georgiadis, MD, Principal Investigator — ProMedica Toledo Hospital
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No